CLINICAL TRIAL: NCT06259994
Title: Obstetrical, Endocrine and Metabolic Consequences of Antenatal Dexamethasone Treatment in Pregnant Women at Risk of Congenital Adrenal Hyperplasia
Brief Title: Dexamethasone and Pregnancy: Maternal Effects
Acronym: DEXAPREG
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231275
Record Dates: First submitted 2024-01-24; First posted 2024-02-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dexamethasone During Pregnancy
Keywords: Congenital Adrenal Hyperplasia 21 hydroxylase pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women treated with dexamethasone during pregnancy at risk of Congenital Adrenal Hyperplasia: All women treated with DEX during pregnancy at risk of Congenital Adrenal Hyperplasia over the defined period (retrospective and prospective).

SUMMARY:
This study will analyze obstetric, endocrine and metabolic follow-up data in women treated with DEX. It will reveal the prevalence and importance of weight gain, insomnia, edema, stretch marks, arterial hypertension and gestational diabetes, describe pregnancy outcome, and analyze the corticotropic axis during and up to 3 months after pregnancy, with the aim of improving the management of these women and preventing comorbidities.

A few studies suggest problems in women treated with DEX during pregnancy. However, all these studies are retrospective, based on self-questionnaires, and have not evaluated all pregnancy outcomes. Moreover, it would appear that a third of women treated with DEX no longer wish to resume the treatment (8). Compliance with treatment is strongly linked to its efficacy. It is therefore important to start investigating the pregnancy outcomes of women treated with DEX. This project is relevant because it has the potential to improve current clinical practice and recommendations related to this treatment, and thus have a direct impact on future patient care. The results of this study will guide us in the management of women presenting an indication for prenatal DEX treatment, and will help to inform the Order of November 15, 2022.

DETAILED DESCRIPTION:
Main objective:

The main aim of this study was to assess the incidence of metabolic complications (hypertension and diabetes) in mothers treated with DEX during pregnancy.

Secondary objectives:

1. To assess the prevalence and importance of adverse effects of DEX: weight gain, stretch marks, insomnia in mothers treated with DEX.
2. Describe pregnancy outcomes and compare them with a reference population (data from the 2010 French perinatal survey (15)).
3. Analyze the corticotropic axis of DEX-treated mothers during and after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Femme majeure (âge ≥ 18 ans)
2. Grossesse avec indication de traitement anténatal par dexaméthasone (DEX) en accord avec le PNDS :

   * Mutation sévère du gène CYP21A2 chez chacun des parents
   * Fœtus féminin
3. Grossesse unique
4. Ayant commencé un traitement anténatal par DEX depuis au moins 24h

Exclusion Criteria:

1. Contraindication to dexamethasone treatment
2. Objection to use of data
3. Persons under legal protection (curatorship, guardianship), court-appointed guardians

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women treated with dexamethasone during pregnancy at risk of Congenital Adrenal Hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who developed hypertension and/or diabetes in mothers treated with DEX | on completion of studies, on average 4 year
  proportion of patients who developed hypertension and/or diabetes in mothers treated with

SECONDARY OUTCOMES:
Assess weight gain, stretch marks and insomnia in mothers treated with DEX Describe complications and illnesses of pregnancy Cortisol and S-DHEA levels during DEX treatment | on completion of studies, on average 4 year
  1. Assess weight gain in kilograms, stretch marks and insomnia in mothers treated with DEX
  2. Describe complications and illnesses of pregnancy, delivery and neonatal outcome: spontaneous or fetal miscarriage, death, hemorrhage in the second or third trimester, or any other medical problem during pregnancy, cesarean section, induced labor, gestational age in days, birth weight in kilograms, etc.
     Compare these data with the outcome of the pregnancy, and with a reference population (data from the 2010 French perinatal survey (15)).
  3. Cortisol and S-DHEA levels during DEX treatment, baseline and regular Synacthen® cortisol levels after DEX discontinuation, duration of hydrocortisone substitution in weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anne BACHELOT, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (17):
- France (17):
  - Hopital Haut Leveque - Endocrinologie, Bordeaux
  - Endocrinologie - Hospices civils de Lyon, Bron
  - Hospices civils de Lyon Biochimie et Biologie moléculaire UM Pathologies endocriniennes, Bron
  - Hospices civils de Lyon Laboratoire de Biologie Médicale Multi Sites, Bron
  - Hospices civils de Lyon Service de médecine de la reproduction, Bron
  - Endocrinologie - CHU Grenoble - Hôpital Michallon, Grenoble
  - Endocrinologie et médecine de la reproduction - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
  - Endocrinologie pédiatrique - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
  - Hopital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille - Hôpital Claude Huriez Endocrinologie, diabétologie et métabolisme, Lille
  - Biologie et médecine de la reproduction, centre d'Assistance Médicale à la Procréation - CHU Nantes - Hôpital Mère et Enfant, Nantes
  - Hospital Saint-Antoine, Endocrinology service, Paris
  - Endocrinologie et médecine de la reproduction-Pitié Salpetriere Hospital, Paris
  - Endocrinologie Pédiatrique-Hôpital Robert Debré, Paris
  - Endocrinologie Pédiatrique-Hôpital Universitaire Necker Enfants Malades, Paris
  - CHU de Toulouse - Hôpita Larrey, Toulouse
  - Pédiatrie - Endocrinologie, génétique et gynécologie médicale - CHU Toulouse - Hôpital des enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No